CLINICAL TRIAL: NCT04311983
Title: Expanding Population-level Interventions to Help More Low-income Smokers Quit
Brief Title: Interventions to Help More Low-income Smokers Quit
Acronym: SFH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202002125-1001; 1R01CA235773-01A1 (NIH); NCT04427839 (obsolete NCT alias)
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Tobacco Use Cessation; Smoking Behaviors; Health Disparity
MeSH Terms: conditions — Tobacco Use Cessation; Smoking

STUDY DESIGN:
Intervention Model Description: Two group intervention; standard care vs. standard + additional service
Who Masked: Participant, Investigator
Masking Description: Participants are unaware of the arms and principal investigators are unaware of participant's randomization to study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tobacco Quitline only (Active Comparator): Smokers in this study group will be offered their state Tobacco Quitline programs
  Interventions: Behavioral: Tobacco Quitline
- Tobacco Quitline plus Smoke Free Homes (Experimental): Smokers in this study group will be offered their state Tobacco Quitline programs, but if they decline, they will be offered a Smoke Free Homes intervention
  Interventions: Behavioral: Tobacco Quitline; Behavioral: Smoke Free Home

INTERVENTIONS:
Behavioral: Tobacco Quitline — Tobacco quitlines provide phone counseling from a quit coach, often supplemented with NRT (nicotine replacement therapy), a quit guide, text messages, or other support. Smokers can call directly or consent to be called by the quitline ("fax-back").
Behavioral: Smoke Free Home — The intervention guides participants though a 5-step process: (1) deciding to create a smoke-free home; (2) talking about it with household members; (3) setting a date for the home to become smoke-free; (4) making the home smoke-free; and (5) keeping the home smoke-free. Progress from one step to the next is facilitated over a 6-week period by three mailings sent to participants' homes and one telephone counseling call delivered by a trained smoke free homes coach.
  Arms: Tobacco Quitline plus Smoke Free Homes

SUMMARY:
In a Hybrid Type 2 randomized trial, 1,980 low-income smokers from nine states with high smoking prevalence will be recruited from 2-1-1 helplines to receive either current standard practice (Quitline) or expanded services (Quitline + Smoke Free Homes) to increase tobacco cessation.

DETAILED DESCRIPTION:
There is an urgent need to engage more low-income smokers in activities that lead to quitting. The current standard of practice for population-level tobacco treatment is phone-based cessation counseling delivered by state tobacco quitlines. But quitline services are restricted to smokers who are ready to quit in the next 30 days, a criterion met by only 20-30% of low-income smokers. Thus, current population level tobacco treatment has nothing to offer 70-80% of low-income U.S. smokers. Based on extensive preliminary research by our study team, the investigators assert that offering a pre-cessation intervention - Smoke Free Homes - to low-income smokers who are not yet ready to quit will: (1) engage more smokers in using proven interventions; (2) increase their readiness to quit and quit attempts; (3) reduce the number of cigarettes they smoke per day; and (4) increase cessation. These benefits will accrue in addition to reducing exposure to harmful secondhand smoke for non-smokers in the home. In a Hybrid Type 2 randomized trial, 1,980 low-income smokers from nine states with high smoking prevalence will be recruited from 2-1-1 helplines to receive either current standard practice (Quitline) or expanded services (Quitline + Smoke Free Homes). In the latter condition, smokers will be offered cessation counseling first, just like current standard practice, but those who decline will then be offered Smoke Free Homes. At 3-month followup, those in the latter condition who accepted quitline services but did not quit will be offered Smoke Free Homes, and those that accepted Smoke Free Homes but did not quit will be offered quitline services. The effectiveness portion of the Hybrid Type 2 design (Aim 1) will use intent-to-treat analyses to compare group differences at 3- and 6-month follow-up in 7- and 30-day point prevalence abstinence with biochemical verification, as well as 24-hour quit attempts and cigarettes smoked per day. The implementation portion of the Hybrid Type 2 design (Aims 2-3) will measure smokers' acceptance and use of the interventions, as well as cost-effectiveness and cost-benefits of adding Smoke Free Homes to quitline services. With rates of smoking and smoking-related cancers much higher in low-income populations and treatment costs exceeding tens of billions of dollars annually in Medicaid alone, this large-scale practical trial will provide strong evidence with high external validity to answer an important policy question: Will changing the standard practice for population-level treatment of smoking result in increased cessation in low-income populations?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21
* English-speaking
* Daily smoker
* Does not have a full home smoking ban
* Recruited from those who called 2-1-1 for themselves and are not in acute crisis

Exclusion Criteria:

-Pregnant women, because recommended tobacco cessation actions differ for this subset of smokers

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1973 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kreuter, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The HCRL Data Center will make the datasets and other materials available without cost to researchers and analysts after a data sharing agreement is completed. Consistent with NIH guidelines, the data sharing agreement: (1) records a request for data use and detailed description of the intent of use; (2) details the study's publication guidelines, including acknowledging and citing project personnel as appropriate; (3) ensures IRB compliance, including not using these data for non-research purposes; and (4) stipulates that users will not share or distribute the data to others without written permission.

REFERENCES:
- [Derived] McQueen A, Wolff J, Grimes L, Teshome E, Garg R, Thompson T, Carpenter K, Kegler MC, Kreuter MW. Comparing acceptance of smoking cessation and smoke-free home intervention offers and associated factors among people with low income in the USA: baseline results of a randomised controlled trial. BMJ Public Health. 2024 Apr 22;2(1):e000843. doi: 10.1136/bmjph-2023-000843. eCollection 2024 Jun. PMID 40018164
- [Derived] Wolff JM, McQueen A, Garg R, Thompson T, Fu Q, Brown DS, Kegler M, Carpenter KM, Kreuter MW. Expanding population-level interventions to help more low-income smokers quit: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2023 Jun;129:107202. doi: 10.1016/j.cct.2023.107202. Epub 2023 Apr 18. PMID 37080354
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tobacco Quitline Only | Tobacco Quitline Plus Smoke Free Homes
Started | 987 | 986
Completed | 558 | 521
Not Completed | 429 | 465
Not completed — Lost to Follow-up | 421 | 456
Not completed — Incomplete survey | 7 | 9
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobacco Quitline Only | Tobacco Quitline Plus Smoke Free Homes | Total
Number analyzed (Participants) | 987 | 986 | 1973
Age, Continuous [Median (Full Range); unit: years] | 51 [21 to 82] | 51 [23 to 85] | 51 [21 to 85]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 317 | 304 | 621
  Female | 665 | 677 | 1342
  Unknown | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 52 | 98
  Not Hispanic or Latino | 939 | 928 | 1867
  Unknown or Not Reported | 2 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 456 | 463 | 919
  Black/African American | 405 | 406 | 811
  American Indian/Alaskan Native | 14 | 17 | 31
  Asian/Asian American | 2 | 0 | 2
  Native Hawaiian/Pacific | 1 | 3 | 4
  Other | 37 | 27 | 64
  Multiracial | 65 | 52 | 117
  Unknown/Missing | 7 | 18 | 25
Region of Enrollment [Number; unit: participants]
  United States | 987 | 986 | 1973

OUTCOME MEASURES:

1. Primary Outcome: 7day Point Prevalence for Smoking
Description: Percentage of participants who have 7 day smoking abstinence
Time Frame: 6 month follow-up
Population: Participants were not included if they were lost to follow-up or were duplicate enrollees.
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Quitline Only | Tobacco Quitline Plus Smoke Free Homes
Number analyzed (Participants) | 560 | 530
Participants | 78 | 83

2. Secondary Outcome: Proportion of Participants Who Accept the Tobacco Quitline Program
Description: * All participants are asked at baseline if they are interested in trying the <STATE> tobacco quitline. Some participants are asked this question again at the 3-month follow-up
  * The probability is the proportion who answer "yes".
  * Due to our study design, at 3-month follow-up, Tobacco Quitline plus Smoke Free Homes participants were only offered the Quitline if they had not chosen it at baseline. The proportion in the table is the number of participants who accepted the Quitline divided by number who were offered the Quitline.
Time Frame: Baseline and 3-month follow-up
Population: At baseline, participants weren't included if they were duplicate entries. At 3-month follow-up, participants weren't included if they were duplicated entries or if they were lost to follow-up. Also, in Arm 2 at 3-month follow-up, if participants had chosen the quitline at baseline and did not quit, they were not re-offered the quitline; they were only offered Smoke-Free Homes. This was a planned part of the study design.
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Quitline Only | Tobacco Quitline Plus Smoke Free Homes
Number analyzed (Participants) | 987 | 986
Participants
  Baseline | 592 | 587
  3-month follow-up: number analyzed (Participants) | 567 | 264
  3-month follow-up | 385 | 142

ADVERSE EVENTS:
Time Frame: From date of enrollment through completion of follow-up (up to 6 months).
Arm/Group | Tobacco Quitline Only | Tobacco Quitline Plus Smoke Free Homes
All-Cause Mortality (participants affected / at risk) | 1/987 | 0/986
Serious Adverse Events (participants affected / at risk) | 0/987 | 0/986
Other Adverse Events (participants affected / at risk) | 0/987 | 0/986

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT04311983/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT04311983/ICF_001.pdf